CLINICAL TRIAL: NCT04551976
Title: Habits of Gamers Study
Acronym: GAMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Gerald Davison, Professor of Psychology, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UP-20-00148
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Depression Mild; Depression, Anxiety; Anxiety; Attention Concentration Difficulty
Keywords: mindfulness
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: 2 x 2 study design with four groups. Half the participants will be randomized to a control condition and half will be randomized to an experimental condition (i.e., mindfulness). All participants will complete each of two study activities, but the order of the activities will be crossed over so that order effects for the activity are minimized. Thus, the groups will be as follows:
  Group 1: mindfulness condition and play video game first, fold laundry second Group 2: mindfulness condition and fold laundry first, play video game second Group 3: control condition and play video game first, fold laundry second Group 4: control condition and fold laundry first, play video game second
Who Masked: Participant
Masking Description: Participants in the control condition are told that we are interested in better understanding the behavioral habits of gamers. We ask them to complete the tasks as they normally would. Every participant will be debriefed after the final study session has concluded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindful Video Game Then Laundry Group (Experimental): Receive mindfulness prompt and play their video game first and fold laundry second.
  Interventions: Behavioral: Mindfulness
- Mindful Laundry Then Video Game Group (Experimental): Receive mindfulness prompt and fold laundry first, play their video game second.
  Interventions: Behavioral: Mindfulness
- Control Video Game Then Laundry Group (No Intervention): Control condition that receives no mindfulness prompt and is asked to complete activities like they normally would. They will play their video game first and fold laundry second.
- Control Laundry Then Video Game Group (No Intervention): Control condition that receives no mindfulness prompt and is asked to complete activities like they normally would. They will fold laundry first and will play their video game second.

INTERVENTIONS:
Behavioral: Mindfulness — Pay attention to the present moment, on purpose, in a nonjudgemental way.
  Arms: Mindful Laundry Then Video Game Group; Mindful Video Game Then Laundry Group

SUMMARY:
Rationale:

Mindfulness is a popular therapeutic strategy that has a growing body of evidence suggesting it can improve a wide range of physical and psychological symptoms. Yet, confusion exists as to why mindfulness is effective as well as the most effective ways in which to teach and practice mindfulness. The present study will test a mindfulness training protocol to better understand the most effective ways to teach and practice mindfulness.

Intervention:

A group of video game players, or "gamers", will be instructed on how to play a video game of their choice in a more mindful way and compare this to an activity of daily functioning (i.e., folding laundry). Outcomes from self-report measures taken both before and after study activities will be tested against a control group of gamers who will perform the same study activities without the mindfulness induction.

Objective or Purpose:

The purpose of the present study is to test the effects of a brief, standardized mindfulness prompt in order to better understand effective ways to train mindfulness concepts. The mindfulness prompt will be applied to an intrinsically motivated activity (i.e., video game play for experienced gamers) and an activity of daily functioning (i.e., laundry folding) in order to evaluate the different effects of mindfulness practice when implemented with a popular leisure activity versus a less engaging activity of daily living.

Study Population:

This study will include adult "gamers" ages 18-65. A gamer is someone who engages in some form of digital video game play for a minimal average of three hours per week. A pre-screening measuring will rule out any participants who do not play video games with enough frequency to be considered a gamer. Study sessions will take place remotely overseen via a Zoom-based video call with study personnel. Another exclusion criteria will be an inability to speak with study personnel via Zoom or do not have a private area to perform the study activities.

Study Methodology:

To address the aims of this study a mixed-method, between- and within-group, counterbalanced study design will be employed. Thus, participants will be randomized to either a mindfulness or control condition with pre- and post-study-task self-report measures collected at two separate study sessions in order to statistically analyze the study hypotheses.

Study Aims:

The present study has one primary aim and several secondary aims: The primary aim is to test the beneficial effects of a standardized, brief mindfulness induction prior to the completion of two different activities (i.e., play a video game or fold laundry). A secondary aim is to evaluate the impact that the type of activity has on one's ability to practice mindfulness. In addition to the primary and secondary aims, an exploratory analysis will be utilized in order to better understand what factors may have mediated the results from the first two aims.

Study Outcomes or Endpoints:

A main effect will be used to test the differences between the study manipulation (i.e., mindfulness prompt) and control (i.e., perform the task as you usually do) conditions. The primary outcome will be a self-reported state-mindfulness scale that measures the degree to which one "mindfully" performed a specific activity. Secondary outcomes will capture changes in emotions from pre- to post-activity, level of engagement or "flow" during the activity, enjoyment performing study activities, and level of focus/concentration during study activities.

Follow-up: No follow-up is planned at this time. A baseline screening measure as well as in-session pre and post-study task questions will be the only data collected.

Statistics and Plans for Analysis:

For the primary aim of the study, a repeated measures multivariate analysis of variance (MANOVA) with a 2 (study group) X 2 (activity type) X 2 (state mindfulness) matrix. The second study aim will be tested with a repeated measures multivariate analysis of covariation (MANCOVA) with the covariates of changes in emotions from pre- to post-activity, level of engagement or "flow" during the activity, enjoyment performing study activities, and level of focus/concentration during study activities.

DETAILED DESCRIPTION:
The present study has been designed to address several shortcomings in the "mindfulness" literature. Mindfulness has been defined as, "paying attention in a particular way: on purpose, in the present moment, and nonjudgmentally." Mindfulness-based interventions have shown an ability to alleviate a wide range of psychological disorders including anxiety and depression and have been integrated into many popular and evidence-based psychotherapeutic modalities including Cognitive Behavioral Therapy (CBT), Dialectical-Behavior Therapy (DBT), and Acceptance and Commitment Therapy (ACT), to name a few. Consequently, a better understanding of the most effective ways to teach mindfulness may help improve the positive effects of existing mindfulness-based interventions and may also inform future intervention and dissemination strategies based on this technique.

One shortcoming of existing mindfulness research is that little consensus exists on how to operationalize the practice of mindfulness and few studies exist in which mindfulness is taught using a brief, standardized method. This is problematic because a lack of such brief and standardized training methods has led to inconsistencies and broad differences in how mindfulness interventions, to date, have defined, operationalized, and applied mindfulness principles and practice strategies. Moreover, it has been suggested that this literature suffers from an over-reliance on long-term, randomized clinical trials, which has resulted in a lack of controlled laboratory-based studies in which the mediating variables responsible for observed changes can be tested. Stated another way, mindfulness lacks research that is controlled, systematic and laboratory-based. Consequently, investigators still understand little about why mindfulness is effective as well as what factors may enhance or hinder one's ability to learn mindfulness strategies. A nebulous understanding of how to operationalize mindfulness and what mechanisms are responsible for change within mindfulness-based interventions should be addressed because the effectiveness of such interventions may be limited and may also lead to misattributions for what factors are mediating the positive effects demonstrated in these interventions. The present study will address this limitation by replicating an existing mindfulness study in which a brief, standardized mindfulness intervention was compared to a control group. The present study will apply similar mindfulness instructions to a different set of activities. This mindfulness manipulation will be compared to a control group receiving no mindfulness instructions.

The first aim of this study, to test a brief, standardized mindfulness prompt prior to the completion of an activity, is meant to address the aforementioned shortcomings in current mindfulness literature. This study will be a partial replication of a systematic investigation conducted by Hanley, who tested a brief, standardized mindfulness induction prior to the completion of an instrumental activity of daily living (i.e., dishwashing) and compared the effects to a control group performing the same activity with no mindfulness prompt. Instrumental activities of daily living like meal preparation, shopping and cleaning are often used to teach mindfulness. Hanley found that participants in the mindfulness condition reported significantly greater levels of mindfulness during the activity, greater levels of positive emotions following the task, more engagement in the activity, and significantly lower levels of negative emotions as compared to the control condition. The present study will employ a similar set of mindfulness instructions prior to the completion of a different activity of instrumental daily living, folding laundry. A similar set of outcomes in relation to state-mindfulness, current emotional states, and experience performing the activity will also be utilized in the present study. This study will be a partial replication and extension of Hanley work. If similar results are observed in the present study it will suggest that brief, standardized mindfulness interventions may be flexibly applied to a wide range of activities. This, in turn, may help increase the opportunities one has to practice mindfulness throughout the day. Consistent practice has been demonstrated to be one of the most important factors in learning mindfulness. Thus, a brief, standardized set of mindfulness instructions that can be flexibly applied to a number of activities may improve the effectiveness of future mindfulness interventions.

The second aim, which is intended to better understand the impact that type of activity has on a mindfulness prompt, may also help further mindfulness literature in several important ways. First, evidence suggests that in addition to consistent practice, feeling engaged and motivated while practicing may also help enhance mindfulness training. By asking participants to complete an activity after receiving mindfulness instructions for both video game play (VGP) and folding laundry the present study will be able to directly compare the differences between mindfulness training when applied to an engaging activity versus a routine activity. VGP was chosen to represent an engaging activity because VGP is a popular global activity that is practiced by millions of people on a daily basis. It has been suggested that VGP may represent an ideal platform in which to teach mindfulness because the real-time feedback and interactivity they provide can keep a user continuously engaged and immersed in the present moment. Much of the engagement and immersion observed during VGP studies may be attributed to the fact that many people find VGP to be a fun, enjoyable, intrinsically motivated activity. Intrinsic motivation, the motivation one feels to engage in activities that they enjoy, has been consistently shown to be one of the most powerful forms of human motivation. Further, people tend to feel the greatest sense of satisfaction and enjoyment when they engage in intrinsically motivated activities. Another reason VGP was selected as an activity for the present study is the emerging body of literature that suggests VGP can act as a platform for psychoeducation and enhance a wide range of behavioral and mental health functions including improved emotion regulation, ability to navigate negative emotions, problem solving, and social interactivity.

In sum, this study is needed in order to better understand optimal ways in which to train and practice mindfulness. More studies like this are needed because the current mindfulness literature lacks systematic investigations of brief, standardized training methods. This has led to a dearth of knowledge about how to operationalize the term "mindfulness" as well as why existing mindfulness interventions have been effective. The present study will address these shortcomings by comparing a brief, standardized mindfulness manipulation when applied to VGP and laundry folding. A between-subjects analysis will be used to test the effects of the mindfulness prompt when compared to a control group. A within-subject analysis will be used to test whether the application of mindfulness to an enjoyable activity (i.e., video game play) produces greater effects than when it is applied to a more routine activity (i.e., folding laundry). This is intended to help inform future mindfulness interventions by providing more insight into effective ways to teach and practice mindfulness.

Risks to participants: This study will present minimal risk to the participants for a variety of reasons. First, a brief screening measure will be used to exclude participants who don't meet our inclusion criteria (including screen out minors). Second, the two study tasks are non-invasive and present no health risks to participants. Specifically, folding laundry and playing a self-selected video game are common activities that participants should be familiar with and that present no inherent dangers to the participants. Third, the questionnaires within the study will be focused on assessing how participants are currently feeling and how they felt about the performance of study task from a variety of questionnaires. Since the questions are tied to a specific task and current thoughts and feelings, they should not present any prompts that participants would find distressing or offensive. Fourth, the mindfulness prompt in this study will be modeled after an existing study which demonstrated effectiveness in teaching participants principles of mindfulness when compared to a control group while also presenting minimal risk to participants. Finally, it will be made clear to participants during the informed consent process that they will be able to leave the study at any time and that they are under no obligation to complete both study sessions. Given these reasons, it is believed the present study does not present any undue risks to participants.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-64
* "Gamer" = must play at least 3 and no more than 30 hours per week
* Must read and speak English
* Must have a private area, of the participant's choosing, in which to complete the two study sessions Must be able to speak with study personnel via Zoom

Exclusion Criteria:

* "Gamer" = less than 3 hours of play per week, or more than 30 hours per week Prior experience with mindfulness in the form of
* "Formal Mindfulness Training". Formal mindfulness training is considered any class, group, or training that was done via individual group psychotherapy, with a licensed mental health professional.
* Be able to fluently read and speak English

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS-X) | Administered prior to the intervention to 10 minutes after the intervention for sessions 1 and 2.
  The Positive and Negative Affect Schedule is a 5-point Likert scale with a minimum value of "1" (very slightly or not at all) and a maximum value of "5" (extremely). The Positive and Negative Affect Schedule measures participants' emotions/affect in the present moment. For this study the Positive and Negative Affect Schedule will be administered prior to and then immediately following a study activity and the change score from pre- to post-activity will constitute a primary outcome. Higher scores on the Positive and Negative Affect Schedule indicates more extreme emotional experiences.
State Mindfulness Scale (SMS) | Administered 15 minutes after the intervention for sessions 1 and 2
  The State Mindfulness Scale is a 5-point Likert scale with a minimum value of "1" (not at all) and a maximum value of "5" (very well). The State Mindfulness Scale measures how "mindfully" one performed a specific task or activity. Higher scores on the State Mindfulness Scale indicate one performed a task in a more mindful way.

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory (IMI) | Administered 20 minutes after the intervention for sessions 1 and 2.
  The Intrinsic Motivation Inventory is a 7-point Likert scale with a minimum value of "1" (not at all) and a maximum value of "7" (extremely true). The Intrinsic Motivation Inventory measures how much enjoyment and satisfaction one derives from engaging in a given activity. Higher scores on the Intrinsic Motivation Inventory indicate more satisfaction and enjoyment for the activity.
Flow State Scale (FSS) | Administered 25 minutes after the intervention for sessions 1 and 2.
  The Flow State Scale is a 5-point Likert scale with a minimum value of "1" (strongly disagree) and a maximum value of "5" (strongly agree). The Flow State Scale measures how immersed one was while performing a task or activity. A higher score on the Flow State Scale indicates that one was more immersed and present during a specified activity.
Qualitative and Quantitative Feedback for Likelihood to Continue Activity in the Future (QQFLCA) | Administered 30 minutes after the intervention for sessions 1 and 2.
  Qualitative and Quantitative Feedback for Likelihood to Continue Activity in the Future are open-ended text-response questions that asks participants for feedback to a variety of questions. The questions ask whether they found the study activity useful and/or important to them.

OTHER OUTCOMES:
Acceptability of mindfulness (AoM) | Administered 45 minutes after the intervention for sessions 1 and 2.
  Acceptability of mindfulness is a multiple choice question that asks participants how easy or difficult they found mindfulness to be, as well as whether it was easier to practice with a video game or via laundry folding. The scale has response options of "video game play," "folding laundry," "both," and "neither."
Semantic Differentiation Scale for Ease of Learning (SDS-EL) | Administered 35 minutes after the intervention for sessions 1 and 2.
  The Semantic Differentiation Scale for Ease of Learning is a semantic differentiation scale with a given a set of word anchors (i.e., happy versus unhappy, pleased versus annoyed, hopeful versus despairing, etc.) that have 7 selection options in between the two words. Participants are asked to place a mark on one of the 7 selection options according to which word better represents how they feel. For data analysis purposes the three selection options closer to a negative word (i.e., unhappy, annoyed, despairing) will be scored -1, -2, and -3 with -3 representing an extreme negative feeling. The three selection options closer to a positive word (i.e., happy, pleased, hopeful) will be scored 1, 2, and 3 with a 3 representing an extreme positive feeling. Selecting a mark in the middle will be scored 0 for neutral. The scale will measure the extent to which participants found the intervention (i.e., mindfulness) to be easy to learn and apply to the study activity.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Davison, Ph.D., Study Chair — Faculty PI
Locations (1):
- Department of Psychology; University of Southern California, Seely G Mudd Building, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson CA, Sakamoto A, Gentile DA, Ihori N, Shibuya A, Yukawa S, Naito M, Kobayashi K. Longitudinal effects of violent video games on aggression in Japan and the United States. Pediatrics. 2008 Nov;122(5):e1067-72. doi: 10.1542/peds.2008-1425. PMID 18977956
- [Background] Baer, R. A. (2003). Mindfulness training as a clinical intervention: A conceptual and empirical review. Clinical psychology: Science and practice, 10(2), 125-143.
- [Background] Baer, R. A. (Ed.). (2015). Mindfulness-based treatment approaches: Clinician's guide to evidence base and applications. Elsevier.
- [Background] Baranowski T, Buday R, Thompson DI, Baranowski J. Playing for real: video games and stories for health-related behavior change. Am J Prev Med. 2008 Jan;34(1):74-82. doi: 10.1016/j.amepre.2007.09.027. PMID 18083454
- [Background] Brown, K. W., Ryan, R. M., & Creswell, J. D. (2007). Mindfulness: Theoretical foundations and evidence for its salutary effects. Psychological inquiry, 18(4), 211-237.
- [Background] Brown, K. W., Ryan, R. M., & Creswell, J. D. (2007). Addressing fundamental questions about mindfulness. Psychological Inquiry, 18(4), 272-281.
- [Background] Gackenbach, J., & Bown, J. (2011). Mindfulness and video game play: A preliminary inquiry. Mindfulness, 2(2), 114-122.
- [Background] Granic I, Lobel A, Engels RC. The benefits of playing video games. Am Psychol. 2014 Jan;69(1):66-78. doi: 10.1037/a0034857. Epub 2013 Dec 2. PMID 24295515
- [Background] Hanley, A. W., Warner, A. R., Dehili, V. M., Canto, A. I., & Garland, E. L. (2014). Washing dishes to wash the dishes: brief instruction in an informal mindfulness practice. Mindfulness, 6(5), 1095-1103.
- [Background] Lippelt DP, Hommel B, Colzato LS. Focused attention, open monitoring and loving kindness meditation: effects on attention, conflict monitoring, and creativity - A review. Front Psychol. 2014 Sep 23;5:1083. doi: 10.3389/fpsyg.2014.01083. eCollection 2014. PMID 25295025
- [Background] Lomas, T., Cartwright, T., Edginton, T., & Ridge, D. (2015). A qualitative analysis of experiential challenges associated with meditation practice. Mindfulness, 6(4), 848-860.
- [Background] Ryan RM, Deci EL. On happiness and human potentials: a review of research on hedonic and eudaimonic well-being. Annu Rev Psychol. 2001;52:141-66. doi: 10.1146/annurev.psych.52.1.141. PMID 11148302
- [Background] Sliwinski, J., Katsikitis, M., & Jones, C. M. (2015, September). Mindful gaming: How digital games can improve mindfulness. In IFIP Conference on Human-Computer Interaction (pp. 167-184). Springer, Cham.
- [Background] Snodgrass JG, Lacy MG, Francois Dengah HJ 2nd, Fagan J, Most DE. Magical flight and monstrous stress: technologies of absorption and mental wellness in Azeroth. Cult Med Psychiatry. 2011 Mar;35(1):26-62. doi: 10.1007/s11013-010-9197-4. PMID 21165683
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637